CLINICAL TRIAL: NCT05691036
Title: Bile Acids Metabolism and Genetic Mutation Profile in the Etiopathogenesis of Intrahepatic Cholestasis of Pregnancy in the Indian Population- A Prospective Study
Brief Title: Bile Acids Metabolism and Genetic Mutation Profile in the ICP in the Indian Population
Acronym: ICP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Madhumita Premkumar, ASSOCIATE PROFESSOR, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 2022-2107
Record Dates: First submitted 2022-08-01; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Intrahepatic Cholestasis of Pregnancy; Genetic Mutation; Health Related Quality of Life
Keywords: Intrahepatic cholestasis of pregnancy; Genetic Mutations in pregnancy associated cholestasis; Pruritus
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Pruritus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 8 mL of blood will be drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with ICP: Case: Pregnant women with consistent pruritus or on medication for pruritus associated with an elevated level of serum transaminase alanine transaminase(ALT)>40 IU/L or aspartate transaminase(AST)>37 IU) and raised serum bile acids ≥10µmol/L will be eligible for the inclusion in the study.
- Pregnant women without ICP: Controls: Healthy pregnant women of the same gestational age with routine physical examinations will be enrolled as a control group.

SUMMARY:
Intrahepatic cholestasis of pregnancy (ICP) is a disorder characterized by itching, elevated fasting serum bile acids ≥10μmol/L (and elevated serum transaminases), with increased risks of perinatal complications, including spontaneous preterm labor, fetal distress, infant respiratory distress syndrome, meconium-stained liquor (MSL), and sudden intrauterine death (IUD). The Incidence of ICP varies from 0.1 to 15.6% of all pregnancies, with the highest cases in Chile, South Asia, America, and Scandinavia. The burden of ICP in India according to various states is as follows Punjab (3.1%), Chandigarh (4.8%), Delhi (0.79%), West Bengal (3.3%), and Lucknow (Uttar Pradesh) (2.8%).

DETAILED DESCRIPTION:
Many physiological, anatomical, and hormonal changes occur in the body during pregnancy to facilitate the best possible growth of the fetus. A functional liver and bile acids (BA) milieu are critical for the development of the fetus, and adverse pregnancy outcomes are possible in women who have primary liver disease. Some pre-existing hepatobiliary diseases may be diagnosed incidentally during pregnancy, such as chronic viral hepatitis. Some common pregnancy-related liver diseases are Intrahepatic Cholestasis of pregnancy (ICP), hemolysis elevated liver enzymes and low platelets (HELLP) syndrome, and acute fatty liver of pregnancy (AFLP). ICP is a cholestatic disorder characterized by (i) pruritus, with onset in the second and third trimester of pregnancy, without any primary skin lesions, (ii) elevated fasting serum bile acids ≥10μmol/L (and elevated serum transaminases), (iii) spontaneous relief of signs and symptoms within two to three weeks after delivery, and (iv) absence of other diseases that cause pruritus and jaundice. Many studies have attempted to associate maternal serum bile acids/ total bile acids with adverse fetal outcomes. ICP is associated with increased risks of perinatal complications, including spontaneous preterm labor, fetal distress, infant respiratory distress syndrome, meconium-stained amniotic fluid, and sudden intrauterine death (IUD). Recent data suggest that women with jaundice had higher rates of prenatal abnormalities than women with just pruritus in ICP. Pruritus can appear as early as seven weeks without causing a rash. Itching is usually noticed early on the palms of the hands and the soles of the feet, although it can occur everywhere on the body. Other symptoms of ICP include dark urine, increased clotting time, fatigue, nausea, loss of appetite, jaundice, and discomfort in the upper right quadrant of the abdomen. It may be mild and tolerable for some patients but may also be very severe and disabling. Women with ICP develop mild jaundice and subclinical steatorrhea. Jaundice typically develops 1 to 4 weeks after the onset of pruritus. Subclinical steatorrhea with fat malabsorption leads to vitamin K deficiency resulting in prolonged prothrombin time and postpartum hemorrhage.

The incidence and prevalence of ICP vary with ethnicity and geography. Ethnic distribution of ICP as Caucasian (53.6%), South Asian (22.6%), African (0.6%), Asian (8.4%), and Australian (3.8%) were noted (8). Among the Asians, Asian of Indian origin 1.24%, Pakistan origin of 1.46%, and whites of 0.62% were found to show Indians and Pakistan origin of Asian have a higher prevalence than whites. Concerning the geographic distribution of ICP, the Incidence of ICP varies from 0.1 to 15.6% of all pregnancies, with the highest cases in Chile, South Asia, America, and Scandinavia. In the case of individual countries such as Chile, 9%, Canada, 0.07%, China, 0.32%, and North California, 1.9% incidence were reported. It is more common in South America as compared to other northern European continents. The incidence of ICP was reported as 0.5-1.5% of pregnancies in Finland. As this study will be done among the Indian population, the burden of ICP in India is reported as Punjab at 3.1%, Chandigarh at 4.8%, Delhi at 0.79%, Nepal at 1.1.5%, West Bengal at 3.3%, Lucknow 2.8%, indicating an urgent need to focus and find out cost-effective and early prognosis and diagnosis of ICP.

ICP is a multifactorial disease interplay between genetic, environmental, and hormonal factors. Common risk factors are the history of oral contraceptive pill (OCP) use, twins, selenium deficiency, genetic transporters defects, and recurrence in the subsequent pregnancy. Patients are usually diagnosed in the second and third trimesters, with increased incidence in winter. Genetic factors contribute as risk factors for ICP including mutation in ATP binding cassette family as ATP binding cassette subfamily B member 4(ABCB4), ATP-binding cassette, sub-family B member 11(ABCB11), ATPase Phospholipid Transporting 8B1(ATP8B1), ATP Binding Cassette Subfamily C Member 2(ABCC2), and tight junction protein 2(TJP2) genes. Bile mainly consists of bile salt, organic anions, electrolytes, phosphatidylcholine, and cholesterol. These components are transported by active process against the concentration gradient by specific transporters such as bile salt export pump (BSEP), Sodium taurocholate co-transporting polypeptide (NTCP), major transporter for the secretion of bile acids from hepatocytes into bile in humans. A study on deoxyribonucleic acid (DNA) of the Italian population with the help of polymerase chain reaction (PCR) and automated sequencing. They found five novel variants of mutation in ABCB4 and ABCB11 and confirmed the statistically significant susceptibility to ICP. Environmental factors associated with ICP include seasonal variation, selenium deficiency, and vitamin D deficiency. Hormonal factors such as estrogen level, sulfated progesterone, intake of oral contraceptive pills, and second-trimester hormonal changes in pregnant women can be attributed as risk factors for ICP. In the urine of pregnant women with ICP, sulfated progesterone correlates with the severity of ICP. Apart from these, other risk factors are responsible for ICP, and they found a statically significant association between pregestational diabetes, tobacco use, history of cholecystectomy, history of ICP in a previous pregnancy, and pregnancy-induced hypertension (PIH).

Placental expression of genes due to placental hypoxia and proteins related to apoptosis, oxidative stress, lipid metabolism, cell proliferation, and immunological response are associated with ICP. Increased total serum BAs and changes in BAs profile reverse the transplacental BA(bile acids) gradient, and increased inflammatory cytokines like interleukin 4(IL4), interleukin 6(IL6), interleukin 12 (IL12), and tumor necrosis factor(TNF) cause respiratory distress in infants and preterm delivery. Immune response, vascular endothelial growth factor(VGEF)signaling pathway, and G-protein-coupled receptor signaling were the most common regulatory genes responsible for inflammatory response, vasculogenesis, and angiogenesis, all essential in ICP pathogenesis. Autotaxin (ATX) is lysophosphatidic acid (LPA) essential for angiogenesis and neuronal development during embryogenesis, cellular motility, proliferation, and lymphocyte homing. ATX levels are reported to be increased during pregnancy and correlate positively with gestational age. LPA and ATX levels were significantly higher in ICP. A large prospective study in Sweden revealed severe perinatal outcomes of ICP as spontaneous preterm labor, asphyxia events, meconium staining of amniotic fluid, and placental and membrane changes did not occur until the level of serum bile acid reached>40umol/L. ICP is a pregnancy-related disorder that is expected to resolve after delivery. However, population-based cohort studies revealed that ICP acts as a risk factor for hepatobiliary disease even after the completion of pregnancy. A significant association between hepatitis C virus (HCV), non-alcoholic liver disease, gallstone, and cholelithiasis, with increased risk of non-alcoholic pancreatitis in women, was observed in women with ICP. A population-based cohort study, with an of 0.32%-0.58% of ICP in Sweden, gives a significant risk association of ICP with gestational diabetes, pre-eclampsia, and a nonsignificant association with postpartum hemorrhage. Total serum bile acids >40mmol/l as severe ICP and associated with increased risk of gestational diabetes mellitus(GDM), pregnancy-induced hypertension(PIH) was reported and managed with ursodeoxycholic acid (UDCA).

Some therapeutic agents such as ursodeoxycholic acid(UDCA), rifampicin, antihistaminic drugs, vitamin K and some topical emollients have been used to alleviate nocturnal pruritus/ pruritus in ICP. Some trials related to reducing the adverse perinatal outcome of ICP were done with the administration of UDCA, dexamethasone, cholestyramine, S-adenosyl methionine(SAMe), plasmapheresis, and fish supplements. UDCA is currently the most effective therapeutic agent used in clinical practice to manage ICP. Several meta-analyses with observational studies or randomized trials have been done on the effectiveness of UDCA, but the results are equivocal. Dexamethasone, rifampicin, SAMe, and cholestyramine also have some roles in the management of ICP. However, reducing pruritus and other adverse perinatal outcomes in pregnancy is unclear. UDCA was effective in improving clinical presentation, normalization of serum profile, and a significant reduction in meconium staining, spontaneous birth, or fetal distress compared to the control/ placebo group. Maternal total serum BAs are significantly associated with reduced infant size and are small for gestational age. Since ICP is the most typical pregnancy-related liver disorder, has multifactorial risk factors, has unclear etiopathogenesis, and results in adverse perinatal outcomes. Pruritus may considerably impair the patient's quality of life as a pregnant woman, causing sleep deprivation and psychological suffering. Only a few studies have been done in India concerning ICP, most of which are related to the reference range of total BAs and the prevalence of ICP. There is no Indian data on how ICP affects the quality of life of a pregnant woman or prospective assessment of genetic risk and bile acid metabolism. So, the aim is to determine the bile acid profile and related metabolites in serum, identify prognostic markers of ICP and assess related risk factors, including the effect of medication and the quality of life of patients with ICP. This research will prospectively evaluate perinatal outcomes and genetic risk factors, which have a bearing on neonatal health. Keeping in mind the symptoms and severity of pruritus, the factors affecting the disease course of pregnant women suffering from ICP will also be evaluated.

ELIGIBILITY:
Inclusion Criteria -

* Age > 21 years with consistent pruritus
* Characterized by consistent pruritus associated with elevated levels of serum transaminases (ALT > 40 U/L or AST > 37 U/L) or raised total serum bile acids (≥ 10 µmol/L)
* Able to understand and comply with the requirements of the study and voluntarily agrees to participate in the study by giving written informed consent before any study-related activity is performed
* Voluntary informed consent to participate until their delivery and also willing to be followed until their delivery
* Agrees to provide information on perinatal and maternal outcomes at or after delivery

Exclusion Criteria:

* Viral and Infectious diseases such as hepatitis B virus (HBV), hepatitis C virus (HCV) related liver disease, Epstein Barr virus (EBV), Cytomegalovirus (CMV), human immunodeficiency virus (HIV) infection) hepatitis C virus (HBV), hepatitis E virus (HEV)
* Primary dermatologic diseases associated with pruritus
* Metabolic diseases (including alcohol abuse)
* Other causes of cholestasis (i.e., primary biliary cholangitis (PBC); primary sclerosing cholangitis (PSC)
* Autoimmune liver disease
* Obstructive biliary diseases
* Cholestatic drug-induced liver injury
* Clinical severe conditions that may affect outcomes include heart failure, renal failure, primary cardiopulmonary diseases
* Twins and triplet pregnancy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women aged more than 21 years.
Study Population: Study Population:
  Group 1: Pregnant women with ICP, n= 75 Cases: Pregnant women with consistent pruritus or on medication for pruritus associated with an elevated level of serum transaminase (ALT>40 IU/L or AST >37 IU) and raised serum bile acids ≥10μmol/L will be eligible for inclusion in the study.
  Group 2: Pregnant women without ICP, n=75 Controls: Healthy pregnant women of the same gestational age with routine physical examinations will be enrolled as a control group.
  Setting: PGIMER (Chandigarh, India)
  Study Centre - Departments of Hepatology/ Obstetrics and Gynaecology, PGIMER, Chandigarh
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The baseline profile of serum bile acids (conjugated and unconjugated) in patients with ICP (Intrahepatic cholestasis of pregnancy) and without ICP. | Day 0
  Bile acids profiling will be accessed by using liquid chromatography combined with mass spectrometry (LC-MS/MS)
Change in the profile of serum bile acids (conjugated and unconjugated) in patients with ICP (Intrahepatic cholestasis of pregnancy) and without ICP. | At delivery
  Bile acids profiling will be accessed by using liquid chromatography combined with mass spectrometry (LC-MS/MS)
Role of ABCB11, ABCB4, and ATP8B1 gene mutations in women with ICP | Day 0
  Targeted Next Generation sequencing will be done at baseline
The HRQOL (Health-related quality of life) in patients with ICP and healthy pregnant women. | Day 0
  Short form (SF) health survey questionnaire will be used to access the quality of life in ICP patients

SECONDARY OUTCOMES:
Determine the risk of labor induction, early termination of pregnancy, and operative delivery in the cohort of women with ICP. | At delivery
  During follow-up, delivery-related details and all the perinatal outcomes will be assessed.
At the baseline visit, measurement of pruritus of the visual analog scale (VAS). | Day 0
  Pruritus will be measured on 0-100mm scale.
Change in pruritus of the visual analog scale (VAS) at delivery. | At delivery
  Pruritus will be measured on 0-100mm scale.
Measurement of fasting bile acids, liver function test(LFT) at baseline in pregnant women with ICP. | Day 0
  Fasting bile acids, liver function test
Change in fasting bile acids, liver function test(LFT) in pregnant women with ICP. | At delivery
  Fasting bile acids and liver function test
Association of ICP with other co-morbid diseases such as pregnancy-induced hypertension, fatty liver of pregnancy, gestational diabetes, etc. | day 0
  Other liver related disease with ICP will be assessed
Pedigree analysis concerning family history of ICP. | Day 0
  ICP is genetic, history of ICP will be assessed among the mother and sister sibling of ICP patients

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- Dr. Madhumita Premkumar, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No